CLINICAL TRIAL: NCT02940730
Title: Evaluation of Intravenous and Intraperitoneal Pharmacokinetics of Dalbavancin in Peritoneal Dialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 16-1355
Record Dates: First submitted 2016-10-13; First posted 2016-10-21 (Estimated); Results first posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-02

CONDITIONS: Infectious Peritonitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dalbavancin via IV (Active Comparator): Dalbavancin will be administered via intravenous administration. Patients will undergo plasma fluid pharmacokinetic sampling for determination of dalbavancin concentrations at time zero, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, at time of volume exchange.
  Interventions: Drug: Dalbavancin via Intravenous Administration
- Dalbavancin via IP (Active Comparator): Dalbavancin will be administered as an intraperitoneal administration. Patients will undergo peritoneal fluid pharmacokinetic sampling for determination of dalbavancin concentrations at time zero, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, at time of volume exchange.
  Interventions: Drug: Dalbavancin via Intraperitoneal Administration

INTERVENTIONS:
Drug: Dalbavancin via Intravenous Administration — Patients will undergo plasma fluid pharmacokinetic sampling for determination of dalbavancin concentrations at time zero, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, at time of volume exchange.
  Arms: Dalbavancin via IV
Drug: Dalbavancin via Intraperitoneal Administration — Patients will undergo peritoneal fluid pharmacokinetic sampling for determination of dalbavancin concentrations at time zero, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, at time of volume exchange.
  Arms: Dalbavancin via IP

SUMMARY:
This study will evaluate the pharmacokinetic properties of dalbavancin when administered as an intravenous infusion and instilled into the peritoneal space in patients who are undergoing peritoneal dialysis. The patients will receive intravenous dalbavancin followed by intensive plasma and peritoneal dialyses fluid sampling. Following a washout phase, the patients will then receive dalbavancin instilled into their peritoneal space followed by the same intensive plasma and peritoneal dialyses fluid sampling.

DETAILED DESCRIPTION:
This study is an open label, cross-over study, evaluating the plasma and peritoneal fluid pharmacokinetics (PK) of dalbavancin after either intravenous or intraperitoneal administration. In the first part of the study, ten patients will be administered dalbavancin on study day 0. Pharmacokinetic analysis will be conducted on days 0, 7, and 14. In the second part of the study, the same 10 patients will cross-over and then be administered dalbavancin on study day 0. Pharmacokinetic analysis will be conducted on days 0, 7, and 14.

Sample Size:

Ten (n=10) patients will be evaluated in this pharmacokinetic evaluation. Since this is a descriptive pharmacokinetic study a sample size calculation was not performed

Plasma and peritoneal fluid sampling:

Dalbavancin will be administered on study day 0. On the intravenous administration day dalbavancin will be administered as a 30-minute intravenous (IV) infusion. On the intraperitoneal administration day, dalbavancin will be administered in the peritoneal dialysis fluid with a 6 hour dwell time. On day 0, patients will undergo plasma and peritoneal fluid pharmacokinetic sampling for determination of dalbavancin concentrations at time zero, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, at time of volume exchange. Patients will be given a specimen collection cup and asked to collect ~30 ml of peritoneal dialysate following scheduled nocturnal dwell approximately 24 hours following the administration of dalbavancin administration. Patients will report for a single PK measurement on study days 7 and 14. (18 total plasma and 18 total peritoneal fluid samples per patient). Blood samples will be drawn from a peripherally inserted intravenous catheter. Peritoneal fluid samples will be drawn from the already placed peritoneal dialysis catheter. Blood samples will be immediately centrifuged at 3000g and plasma and peritoneal fluid samples will be stored at -80°C until analysis.

Description, Risks and Justification of Procedures and Data Collection Tools:

Visit 1 and 4: (~8 hours): On visits 1 and 4 the patients will undergo intensive PK sampling. Subjects will be admitted to the Clinical and Translational Research Center (CTRC) in the morning and a "saline-lock" will be placed. A pre-dose sample and safety labs (comprehensive metabolic panel and urine pregnancy test for women of childbearing potential) will be obtained. The dalbavancin 1500 mg will either be administered intravenously (Visit 1) or into the intraperitoneal space (Visit 4) using the patient's existing peritoneal dialysis catheter with the patients currently prescribed dialysate. Following the blood and peritoneal fluid collection at the second dialysis volume exchange, the subjects will be discharged and asked to return at a scheduled time on day 7. Patients will also be given a specimen collection up with instructions to collect approximately 30 ml of peritoneal dialysate following their evening nocturnal dwell. The collected dialysate will be returned to the investigators.

Visit 2, 3, 5, and 6: (~60 minutes): A "saline-lock" will be placed and blood and peritoneal fluid sample will be collected at each of these visits. All blood and peritoneal fluid draws will be completed at the CTRC. The patient will be discharged and follow up visits will be scheduled for day 14 or next intensive PK sampling visit.

Washout: During the washout portion of this study the patients will not be asked to come in for any visits. This time-frame is to ensure that all of the medication (dalbavancin) has left the patients' system before administering another dose of the medication.

Laboratory tests: The laboratory tests to be performed as part of this study include pregnancy testing to confirm eligibility and comprehensive metabolic panels to determine eligibility and evaluate safety.

Pharmacokinetic Assessments: 4 mL of blood will be collected in a purple top (Ethylenediaminetetraacetic acid) tube and 4 mL of peritoneal fluid in a urine collection cup at pre-dose, and 1, 2, 3, 4, 6, dialysis volume exchange 1, 8, dialysis volume exchange 2 post dose for quantification of dalbavancin. Blood and peritoneal fluid will be placed in an ice bath to chill until centrifuged. Plasma will be harvested within 30 minutes of each blood sample and will be stored at -80ºC until assaying.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 to ≤89 years of age
* Actively receiving chronic peritoneal dialysis
* Ability and willingness to provide written informed consent

Exclusion Criteria:

* Patients currently receiving antimicrobial therapy or have received antibiotic therapy within 14 days prior to study
* Patients with known hypersensitivity reactions to dalbavancin or other glycopeptides
* Prisoners
* Pregnant or breastfeeding women
* Decisionally challenged patients

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2018-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ty H Kiser, PharmD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 10 patients were recruited for this study. All patients started in the intravenous therapy arm. After the washout period patients could start the intraperitoneal treatment arm.
Pre-assignment Details: This is a cross-over study. IP arm was stopped after first 3 patients.
Groups:
- Dalbavancin Via IV, Then Via IP: Dalbavancin will be administered via intravenous administration. Patients will undergo plasma fluid pharmacokinetic sampling for determination of dalbavancin concentrations at time zero, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, at time of volume exchange.
  Dalbavancin via Intravenous Administration: Patients will undergo plasma fluid pharmacokinetic sampling for determination of dalbavancin concentrations at time zero, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, at time of volume exchange.
  Dalbavancin via Intraperitoneal Administration: Patients will undergo peritoneal fluid pharmacokinetic sampling for determination of dalbavancin concentrations at time zero, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, at time of volume exchange.
- Dalbavancin Via IP, Then Via IV: Dalbavancin will be administered as an intraperitoneal administration. Patients will undergo peritoneal fluid pharmacokinetic sampling for determination of dalbavancin concentrations at time zero, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, at time of volume exchange.
  Dalbavancin via Intraperitoneal Administration: Patients will undergo peritoneal fluid pharmacokinetic sampling for determination of dalbavancin concentrations at time zero, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, at time of volume exchange.
  Dalbavancin via Intravenous Administration: Patients will undergo plasma fluid pharmacokinetic sampling for determination of dalbavancin concentrations at time zero, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, at time of volume exchange.
Period: Intervention 1
Arm/Group | Dalbavancin Via IV, Then Via IP | Dalbavancin Via IP, Then Via IV
Started | 10 | 0
Received Intervention | 10 | 0
Completed | 10 | 0
Not Completed | 0 | 0
Period: Intervention 2
Arm/Group | Dalbavancin Via IV, Then Via IP | Dalbavancin Via IP, Then Via IV
Started | 10 | 0
Received Intervention | 3 | 0
Completed | 3 | 0
Not Completed | 7 | 0
Not completed — Physician Decision | 7 | 0

BASELINE CHARACTERISTICS:
Population: Because the study was terminated early, no participants were assigned to the Dalbavancin Via IP, Then Via IV arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dalbavancin Via IV, Then Via IP | Dalbavancin Via IP, Then Via IV | Total
Number analyzed (Participants) | 10 | 0 | 10
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55.5 [36 to 68] |  | 55.5 [36 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 |  | 5
  Male | 5 |  | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 7 |  | 7
  More than one race | 3 |  | 3
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants] — Colorado
  participants
    United States | 10 |  | 10

OUTCOME MEASURES:

1. Primary Outcome: Determine Dalbavancin Plasma Area Under the Curve in Peritoneal Dialysis Patients After Intravenous and Intraperitoneal Administration
Description: 14 day plasma concentrations
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: mg*h/L
Arm/Group | Dalbavancin Via IV | Dalbavancin Via IP
Number analyzed (Participants) | 10 | 3
mg*h/L | 40573.2 (9800.3) | 13532.3 (4913.4)

2. Primary Outcome: Determine Dalbavancin Peritoneal Fluid Area Under the Curve in Peritoneal Dialysis Patients After Intravenous and Intraperitoneal Administration
Description: 14 day peritoneal fluid concentrations
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: mg*h/L
Arm/Group | Dalbavancin Via IV | Dalbavancin Via IP
Number analyzed (Participants) | 10 | 3
mg*h/L | 2125 (1794.3) | 69654.3 (55486.5)

3. Secondary Outcome: Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug, Graded According to NCI CTCAE Version 3.0
Description: Adverse reactions
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dalbavancin Via IV | Dalbavancin Via IP
Number analyzed (Participants) | 10 | 3
Participants | 0 | 3

4. Secondary Outcome: Determine Dalbavancin Plasma Clearance in Peritoneal Dialysis Patients After Intravenous and Intraperitoneal Administration
Description: Dalbavancin plasma clearance
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Dalbavancin Via IV | Dalbavancin Via IP
Number analyzed (Participants) | 10 | 3
L/h | 0.0298 (0.00765) | 0.059 (0.039)

5. Secondary Outcome: Determine Dalbavancin Peritoneal Fluid Clearance in Peritoneal Dialysis Patients After Intravenous and Intraperitoneal Administration
Description: Dalbavancin peritoneal fluid clearance
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Dalbavancin Via IV | Dalbavancin Via IP
Number analyzed (Participants) | 10 | 3
L/h | 0.586 (0.192) | 0.034 (0.027)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Dalbavancin Via IV | Dalbavancin Via IP
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/10 | 3/3
Other Adverse Events (participants affected / at risk) | 0/10 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalbavancin Via IV (N=10) | Dalbavancin Via IP (N=3)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 3 (3) — Abdominal Pain with severe bloating

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT02940730/Prot_SAP_000.pdf